CLINICAL TRIAL: NCT03999515
Title: Erdafitinib Plus Abiraterone Acetate or Enzalutamide in Double Negative Prostate Cancer
Brief Title: Erdafitinib and Abiraterone Acetate or Enzalutamide in Treating Patients With Double Negative Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual
Sponsor: University of Washington (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Principal Investigator, Michael Schweizer, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1005038; NCI-2019-03812 (Registry Identifier: NCI / CTRP); 10288 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-06-21; First posted 2019-06-26 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Castration-Resistant Prostate Carcinoma; Double-Negative Prostate Carcinoma; Metastatic Prostate Carcinoma; Prostate Adenocarcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
Keywords: Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Acetates; Esters; enzalutamide; benzamide; erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (abiraterone acetate, enzalutamide, erdafitinib) (Experimental): Patients receive abiraterone acetate orally PO QD or enzalutamide PO QD on days 1-21. Patients also receive erdafitinib PO QD on days 1-21. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abiraterone Acetate; Drug: Enzalutamide; Drug: Erdafitinib

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: 154229-18-2; 17-(3-Pyridyl)-5; 16-androstadien-3beta-acetate; Androsta-5,16-dien-3-ol; 17-(3-pyridinyl)-; acetate (ester); CB7630; Yonsa; Zytiga; BR9004; BR9004-1; JNJ-212082
Drug: Enzalutamide — Given PO
  Other Names: 915087-33-1; ASP9785; Benzamide; MDV3100; Xtandi
Drug: Erdafitinib — Given PO
  Other Names: Balversa; JNJ-42756493

SUMMARY:
This phase II trial studies how well erdafitinib in combination with abiraterone acetate or enzalutamide works in treating patients with double negative prostate cancer. Erdafitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Testosterone can cause the growth of prostate cancer cells. Abiraterone acetate lowers the amount of testosterone made by the body. This may help stop the growth of tumor cells that need testosterone to grow. Enzalutamide blocks the use of testosterone by the tumor cells. Giving erdafitinib with abiraterone acetate or enzalutamide may work better in treating patients with prostate cancer compared to abiraterone acetate or enzalutamide alone.

DETAILED DESCRIPTION:
OUTLINE: Patients receive abiraterone acetate orally (PO) once daily (QD) or enzalutamide PO QD on days 1-21. Patients also receive erdafitinib PO QD on days 1-21. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 18 years of age prior to signing informed consent
* History of histologically diagnosed prostatic adenocarcinoma
* Participants must have evidence of castration resistant prostate cancer as evidenced by a confirmed rising PSA or radiographic progression (per Prostate Cancer Working Group 3 [PCWG3] criteria) and a castrate serum testosterone level (i.e. =< 50 mg/dL)
* Participants must have previously progressed on abiraterone acetate and/or enzalutamide, with PSA or radiographic progression on the most recent agent per PCWG3 criteria. If the most recent agent received was abiraterone or enzalutamide there should be no washout prior to initiating erdafitinib per protocol
* Measurable disease as defined per RECIST v1.1 criteria
* Subjects who have progressed on only one next-generation AR-directed therapy (e.g. abiraterone, enzalutamide) and who have not received taxane chemotherapy will be required to have evidence of double-negative prostate cancer as defined by immunohistochemistry on biopsy. A fresh metastatic biopsy within 8 weeks is preferred; however, any archival tissue showing a DNPC phenotype will be acceptable for determining eligibility. Patients who have received two prior lines of AR-directed therapy and at least one prior taxane do not require histologic confirmation of DNPC. Note: transcript profiling methods for defining DNPC may be accepted per the PI's discretion
* Eastern Cooperative Oncology Group (ECOG) performance status score =< 2
* Hemoglobin >= 8 g/dL (>= 5 mmol/L) (must be without red blood cell [RBC] transfusion within 7 days prior to the laboratory test)
* Platelets >= 75 x 10^9/L
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (prior growth factor support is permitted but must be without support in the 7 days prior to the laboratory test)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN) or =< 5 x ULN for subjects with liver metastases
* Creatinine clearance >= 40 mL/min/1.73 m^2 based upon modified diet in renal disease formula calculation
* Total bilirubin =< 1.5 x ULN; except in subjects with congenital bilirubinemia, such as Gilbert syndrome
* Corrected QT interval (corrected QT interval by Fridericia [QTcF] or QT corrected interval by the Bazett's formula [QTcB]) =< 480 msec based on the average of triplicate assessments performed approximately 5 minutes apart
* Subjects must agree to use acceptable contraception
* Must sign an informed consent form (ICF) (or their legally acceptable representative must sign) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 14 days prior to randomization
* Active malignancies (i.e., requiring treatment change in the last 24 months) other than malignancy under study (except skin cancers within the last 24 months that is considered completely cured)
* Evidence of predominant small cell or neuroendocrine variant prostate cancer on most recent standard of care metastatic biopsy
* Symptomatic central nervous system (CNS) metastases. Treated CNS metastases will be allowed if these are stable for at least 8 weeks prior to enrollment
* Received prior FGFR inhibitor treatment or if the subject has known allergies, hypersensitivity, or intolerance to erdafitinib or its excipients
* Current central serous retinopathy (CSR) or retinal pigment epithelial detachment of any grade
* Has persistent phosphate level > ULN during screening (on 2 consecutive assessments at least 1 week apart, within 14 days of treatment and prior to cycle 1 day 1) and despite medical management
* Has a history of or current uncontrolled cardiovascular disease including:

  * Unstable angina, myocardial infarction, ventricular fibrillation, Torsades de Pointes, cardiac arrest, or known congestive heart failure class III-V within the preceding 3 months; cerebrovascular accident or transient ischemic attack within the preceding 3 months
  * Pulmonary embolism or other VTE (venous thromboembolism) within the preceding 2 months
* Has known active acquired immune deficiency syndrome (AIDS) (human immunodeficiency virus [HIV] infection)
* Hepatitis B infection as defined according to the American Society of Clinical Oncology guidelines. In the event the infection status is unclear, quantitative levels are necessary to determine the infection status. Hepatitis C (anti-hepatitis C virus [HCV] antibody positive or HCV-ribonucleic acid [RNA] quantitation positive) or known to have a history of hepatitis C. If positive, further testing of quantitative levels to rule out positivity is required
* Has not recovered from reversible toxicity of prior anticancer therapy (except toxicities which are not clinically significant such as alopecia, skin discoloration, hot flashes, grade 1 neuropathy, grade 1-2 hearing loss)
* Has impaired wound healing capacity defined as skin/decubitus ulcers, chronic leg ulcers, known gastric ulcers, or unhealed incisions
* Major surgery within 2 weeks of the first dose, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study or within 2 weeks after the last dose of study drug administration. (Note: subjects with planned surgical procedures to be conducted under local anesthesia may participate
* Any serious underlying medical condition, such as:

  * Evidence of serious active viral, bacterial, or uncontrolled systemic fungal infection
  * Active autoimmune disease or a documented history of autoimmune disease
  * Psychiatric conditions (e.g., alcohol or drug abuse), dementia, or altered mental status
* Any other issue that would impair the ability of the subject to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Patient, who, in the opinion of their treating physician, requires immediate treatment (e.g. those with extensive liver metastases)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schweizer, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Abiraterone Acetate, Enzalutamide, Erdafitinib)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Abiraterone Acetate, Enzalutamide, Erdafitinib)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non Hispanic | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Will be calculated as the percentage of patients, with 95% confidence intervals, achieving a complete response or partial response across the entire study population at any time.
Time Frame: Up to 67 days
Population: Enrolled patients who had re-staging scans performed. Note, study was terminated early due to low accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Abiraterone Acetate, Enzalutamide, Erdafitinib)
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Radiographic Progression Free Survival (PFS)
Description: Progression free survival is time to progressive disease. Disease progression is determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for soft tissue metastases and Prostate Cancer Working Group 3 criteria for bone metastases. Median progression free survival will be calculated.
Time Frame: Up to 67 days
Population: Enrolled patients who had re-staging scans performed. Note, study was terminated early due to low accrual.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Abiraterone Acetate, Enzalutamide, Erdafitinib)
Number analyzed (Participants) | 2
days | 59 [59 to 67]

3. Secondary Outcome: Time to Response
Description: Time to response is the time until a radiographic response occures as determined by RECIST 1.1 criteria. This cannot be determined since only two patients had re-staging scans on study and neither had a response.
Time Frame: Up to 67 days
Population: Enrolled patients who had re-staging scans performed. Note, study was terminated early due to low accrual.
Measure: Number; unit: years
Arm/Group | Treatment (Abiraterone Acetate, Enzalutamide, Erdafitinib)
Number analyzed (Participants) | 2
years | NA — 0 patients achieved a response and therefore time to response cannot be calculated.

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is time to death from any cause. Median overall survival survival will be calculated.
Time Frame: From cycle 1, day 1 to the date of death, assessed up to 178 days
Population: Note, study was terminated early due to low accrual.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Abiraterone Acetate, Enzalutamide, Erdafitinib)
Number analyzed (Participants) | 3
days | 94 [40 to 178]

5. Secondary Outcome: Prostate-specific Antigen (PSA) Response
Description: PSA response will be defined by a > 50% reduction in PSA compared with baseline at any point during treatment. We will report the percentage of patients who achieve a PSA response.
Time Frame: Baseline up to 73 days
Population: Enrolled patients who had repeat PSA performed while on study. Note, study was terminated early due to low accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Abiraterone Acetate, Enzalutamide, Erdafitinib)
Number analyzed (Participants) | 2
Participants | 0

6. Secondary Outcome: Incidence and Severity of Adverse Events (AEs)
Description: Will be assessed using version National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Will characterize AEs by type and grade. Safety will be summarized as the severity and frequency of a given AE.
Time Frame: Within 14 days of end of treatment, an average of 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Abiraterone Acetate, Enzalutamide, Erdafitinib)
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: Within 14 days of end of treatment, an average of 1 year
Arm/Group | Treatment (Abiraterone Acetate, Enzalutamide, Erdafitinib)
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Abiraterone Acetate, Enzalutamide, Erdafitinib) (N=3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Abiraterone Acetate, Enzalutamide, Erdafitinib) (N=3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Dry Eye (Eye disorders) | 1 (1)
Fatigue (General disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight Loss (Investigations) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1)
Nail Changes (General disorders) | 1 (1)
Mouth Sores (General disorders) | 1 (1)
Decreased Appetite (General disorders) | 1 (1)
Nasal Dryness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT03999515/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT03999515/ICF_001.pdf